CLINICAL TRIAL: NCT06281535
Title: Early Versus Conventional Loading for Fully Guided Immediate Implant Placement in Molar Sites (A Randomized Controlled Clinical Study)
Brief Title: Early Versus Conventional Loading for Fully Guided Immediate Implant Placement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Adel Salah Khattab, Associate Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21789
Record Dates: First submitted 2024-02-06; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Dental Implant
Keywords: early loading; conventional loading
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early loading group (Experimental): The surgical treatment protocol entails atraumatic tooth extraction, fixture insertion and placement of the final restoration 2 months following implant placement.
  Interventions: Device: Implant loading
- Conventional loading group (Active Comparator): The surgical treatment protocol entails atraumatic tooth extraction, fixture insertion and placement of the final restoration 3 months following implant placement.
  Interventions: Device: Implant loading

INTERVENTIONS:
Device: Implant loading — Placement of abutments and final restorations either 2 months following implant placement in early loading group or 3 months in conventional loading group

SUMMARY:
Conventional loading protocol following implant placement 3 -6 months is considered the gold standard. However, early loading following 2 months after implant placement decreases the time and had a good survival rate.

DETAILED DESCRIPTION:
The conventional loading protocol presented involves healing period of 3 -6 months. A healing period without stress was recommended in the order to present better survival rate. This loading protocol was developed in the time when micro- and macro design of implant surface was machine produced. Early loading of dental implants within 2 months following placement on healed posterior mandible showed 100% survival rate for five years follow up, with uneventful crestal bone loss. The lack of difference between conventional loading 6 months following implant placement and early loading could be explained by the fact that even if the crowns were not put in direct occlusion, patients used them functionally when chewing. The most relevant factor which may explain the positive results obtained in this trial is the high insertion torque at implant placement.

ELIGIBILITY:
Inclusion Criteria:

* Patients age range from 20-60 years.
* Molar tooth to be extracted due to periodontal diseases, peri- apical diseases, Endo-perio diseases, or tooth fracture.
* Primary implant stability is above 30 Ncm.

Exclusion Criteria:

* History or presence of severe uncontrolled systemic disease.
* Heavy smokers (>10 cigarettes per day) or alcohol/drug abusers.
* Poor oral hygiene.
* Acute periapical infection.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-02-20 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Implant stability | 2 and 3 months following implant placement
  Degree of implant stability will be measured by Osstell device as a scale from 1 to 100

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Adel-Khattab, PhD, Study Chair — Associate Professor Faculty of Dentistry, Ain Shams University; Abdel Rahman Khalaf, PhD, Principal Investigator — Lecturer of Faculty of Dentistry, Assiut University

IPD SHARING:
Plan to Share IPD: No